CLINICAL TRIAL: NCT03870295
Title: Assessment of a New Measurement Technique for Type C Fibre Nerve Conduction Velocity in Polyneuropathies.
Brief Title: Technique to Measure Type C Fibre Nerve Conduction Velocitynerve Fibers in Polyneuropathies
Acronym: FIBREC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Intercommunal de Toulon La Seyne sur Mer (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2018-CHITS-03; 2018-A02621-54 (Other: Id-RCB)
Record Dates: First submitted 2019-03-08; First posted 2019-03-12 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2022-10

CONDITIONS: Peripheral Nervous System Diseases
Keywords: Type C nerve fibres; Conduction velocity; Polyneuropathy
MeSH Terms: conditions — Peripheral Nervous System Diseases; Polyneuropathies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients suffering from polyneuropathies (Experimental): Type C fibre conduction velocity determination in patients suffering from polyneuropathy
  Interventions: Diagnostic Test: Sympathetic skin response (SSR) measure
- Control patients (Active Comparator): Type C fibre conduction velocity determination in control patients
  Interventions: Diagnostic Test: Sympathetic skin response (SSR) measure

INTERVENTIONS:
Diagnostic Test: Sympathetic skin response (SSR) measure — Ankle - ground distance measurement, hand and foot cutaneous temperature reading, low intensity electrical stimulations on hand and on foot to determine SSR at these two points and DN4 questionnaire to assess the possible presence of neuropathic pain

SUMMARY:
Peripheral nerve diseases can separately affect different kind of nerve fibres. Globally two kinds of fibres can be distinguished: large size and small size. The usual electromyogram only investigates large size fibres. Techniques to explore small size fibre function exist but are not used in common practice because of their very specialized aspect or their lack of diagnostic value. The purpose of this study is to develop a measurement technique of small size type C nerve fibre conduction velocity, to show that this velocity is reduced in patients suffering from polyneuropathies and to establish reference values in healthy patients.

DETAILED DESCRIPTION:
Sympathetic skin response (SSR) is one of the simplest means to register the electrophysiological activity of small size nerve fibres. It corresponds to the emission of an electrical potential by sweat glands due to stimulation by type C nerve fibres. These fibres belong to vegetative and somatic nervous systems which can be activated by various stimuli.

Medical applications were considered in the context of polyneuropathies with dysautonomia but SSR did not yield a satisfactory diagnostic value. Parameters used were SSR latency and amplitude. Latency showed little variation with pathology and it is considered that as long as fibres are present their conduction velocity is respected as an all-or-nothing phenomenon. On the contrary, amplitude is very variable, in particular between subjects, which prevents from applying a confidence interval to a given subject. Only unilateral suppression of the response seems to be a reliable criterion and gave results in the context of peripheral nervous pathologies.

The good results obtained with "response suppression" shows SSR sensibility. The discredit of "conduction velocity" variable seems to come from a publication using microneurography. However with this technique only one fascicle is investigated and preferably one giving a good signal, so not representative of all nerve fibres.

Consistent results were achieved with a technique consisting in recording SSR at two points of a same path, separated by a known distance. Knowing the difference of response latency at these two points, velocity could be deduced on the path. This technique was tested in healthy patients in 1988 taking as measurement sites the hand stuck on the body and the ground as a reference for foot plantar. It gave a velocity equivalent to the result found by another team with the same method. The purpose of the study is to apply this technique to pathology.

It should be noted that the velocity measured in this way depends on superior and inferior limb paths, on a medullar portion between C7 et D12 and on pre-ganglionic neurone portion. It has consequently no lesion focalisation capacities and is more appropriate for polyneuropathies with diffuse damage. Nevertheless, it has two advantages. First sweet follicles are in the same functional state in hand and on foot since stimulation intervals are the same at both levels. Secondly the influence of cerebral trunk centres on SSR emission and latency may be bypassed. Thus the study hypothesis is that conduction velocity determination of SSR constituting fibres will better characterize their functional state than response latency measurement which is subject to central excitability variations.

ELIGIBILITY:
Inclusion Criteria for experimental group:

* Patients with polyneuropathy explicit suspicion or whose symptomatology evokes this disease confirmed by electromyogram
* Free informed consent of patient

Inclusion Criteria for control group:

* Patients having a consultation scheduled in neurology department
* Free informed consent of patient

Exclusion Criteria for experimental group:

* Age < 18 years old
* Signs or medical history of central nervous system damage
* Person suffering from another peripheral nervous system pathology than polyneuropathy
* Known or suspected pregnancy and breastfeeding women
* Patients not covered by a social security regimen
* Patients under legal guardianship
* Patients deprived of their liberty due to judicial or administrative decision

Exclusion Criteria for control group:

* Age < 18 years old
* Polyneuropathy suspicion
* Signs or medical history of peripheral or central nervous system damage
* Known or suspected pregnancy and breastfeeding women
* Patients not covered by a social security regimen
* Patients under legal guardianship
* Patients deprived of their liberty due to judicial or administrative decision

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2019-09-30 (Actual); Primary Completion 2020-09-29 (Actual); Study Completion 2020-09-29 (Actual)

PRIMARY OUTCOMES:
Measurement of sudomotor fibre conduction velocity | 30 minutes
  Sudomotor fibre conduction velocity measurement and comparison between patients suffering from polyneuropathy and control patients

SECONDARY OUTCOMES:
Link between neuropathic pain and conduction velocity | 30 minutes
  Correlation between DN4 questionnaire score and conduction velocity

CONTACTS AND LOCATIONS:
Overall Officials: Jacques Grapperon, MD, Study Director — Centre Hospitalier Intercommunal Toulon La Seyne sur Mer
Locations (1):
- Centre hospitalier intercommunal de Toulon La Seyne sur Mer, Toulon, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Arunodaya GR, Taly AB, Swamy HS. Sympathetic skin response in acute sensory ataxic neuropathy. J Neurol Sci. 1995 May;130(1):35-8. doi: 10.1016/0022-510x(94)00271-o. PMID 7650529
- [Background] Vetrugno R, Liguori R, Cortelli P, Montagna P. Sympathetic skin response: basic mechanisms and clinical applications. Clin Auton Res. 2003 Aug;13(4):256-70. doi: 10.1007/s10286-003-0107-5. PMID 12955550
- [Background] Fagius J, Wallin BG. Sympathetic reflex latencies and conduction velocities in normal man. J Neurol Sci. 1980 Sep;47(3):433-48. doi: 10.1016/0022-510x(80)90098-2. PMID 7420119
- [Background] Fagius J, Wallin BG. Sympathetic reflex latencies and conduction velocities in patients with polyneuropathy. J Neurol Sci. 1980 Sep;47(3):449-61. doi: 10.1016/0022-510x(80)90099-4. PMID 7420120
- [Background] Tzeng SS, Wu ZA, Chu FL. The latencies of sympathetic skin responses. Eur Neurol. 1993;33(1):65-8. doi: 10.1159/000116904. PMID 8440291
- [Background] Soliven B, Maselli R, Jaspan J, Green A, Graziano H, Petersen M, Spire JP. Sympathetic skin response in diabetic neuropathy. Muscle Nerve. 1987 Oct;10(8):711-6. doi: 10.1002/mus.880100806. PMID 2825012
- [Background] Valls-Sole J, Monforte R, Estruch R. Abnormal sympathetic skin response in alcoholic subjects. J Neurol Sci. 1991 Apr;102(2):233-7. doi: 10.1016/0022-510x(91)90074-h. PMID 1649263
- [Background] Montagna P, Marchello L, Plasmati R, Ferlini A, Patrosso MC, Salvi F. Electromyographic findings in transthyretin (TTR)-related familial amyloid polyneuropathy (FAP). Electroencephalogr Clin Neurophysiol. 1996 Oct;101(5):423-30. PMID 8913196
- [Background] Carmichael EA, Honeyman WM, Kolb LC, Stewart WK. Peripheral conduction rate in the sympathetic nervous system of man. J Physiol. 1941 Mar 25;99(3):338-43. doi: 10.1113/jphysiol.1941.sp003905. No abstract available. PMID 16995255
- [Background] Sourek K. [Reflex skin potential reactions in cases of surgically tested discopathies]. Acta Univ Carol Med (Praha). 1965:Suppl 21:99+. No abstract available. Multiple languages. PMID 5880965
- [Background] Uncini A, Pullman SL, Lovelace RE, Gambi D. The sympathetic skin response: normal values, elucidation of afferent components and application limits. J Neurol Sci. 1988 Nov;87(2-3):299-306. doi: 10.1016/0022-510x(88)90254-7. PMID 2850351
- [Background] Knezevic W, Bajada S. Peripheral autonomic surface potential. A quantitative technique for recording sympathetic conduction in man. J Neurol Sci. 1985 Feb;67(2):239-51. doi: 10.1016/0022-510x(85)90120-0. PMID 3981220
- [Background] Elie B, Guiheneuc P. Sympathetic skin response: normal results in different experimental conditions. Electroencephalogr Clin Neurophysiol. 1990 Sep;76(3):258-67. doi: 10.1016/0013-4694(90)90020-k. PMID 1697257
- [Background] Sequeira H, Hot P, Silvert L, Delplanque S. Electrical autonomic correlates of emotion. Int J Psychophysiol. 2009 Jan;71(1):50-6. doi: 10.1016/j.ijpsycho.2008.07.009. Epub 2008 Jul 23. PMID 18723054